CLINICAL TRIAL: NCT06397313
Title: An Open-Label Clinical Trial of RVU120 as Monotherapy and in Combination With Ruxolitinib in Patients With Intermediate or High-Risk, Primary or Secondary Myelofibrosis (POTAMI-61)
Brief Title: RVU120 in Patients With Intermediate or High-risk, Primary or Secondary Myelofibrosis
Acronym: POTAMI-61
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ryvu Therapeutics SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POTAMI-61
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Myelofibrosis
Keywords: intermediate; high-risk; primary; secondary
MeSH Terms: conditions — Primary Myelofibrosis; Neoplasm Metastasis | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RVU120 (Experimental): Cohort 1 RVU120 is administered at 250 mg as a single agent every other day on days 1, 3, 5, 7, 9, 11, and 13 of 21-day treatment cycles, or at an adjusted dose, to participants with intermediate or high-risk, primary or secondary MF who have been previously treated with or are ineligible for treatment with a JAK inhibitor.
  Interventions: Drug: RVU120
- RVU120 + ruxolitinib (Experimental): Cohort 2 RVU120 is administered at 250 mg every other day on days 1, 3, 5, 7, 9, 11, and 13 of 21-day treatment cycles or at an adjusted dose, in combined with ruxolitinib administered orally twice daily following the dosing instructions in current prescribing information, to participants with intermediate or high risk, primary or secondary MF experiencing suboptimal response to JAK inhibitor.
  Interventions: Drug: RVU120; Drug: Ruxolitinib

INTERVENTIONS:
Drug: RVU120 — RVU120 is a potent, selective inhibitor of CDK8 and its paralog CDK19
  Other Names: SEL120
Drug: Ruxolitinib — Ruxolitinib is a kinase inhibitor which inhibits Janus Associated Kinases (JAKs) JAK1 and JAK2
  Other Names: RUX
  Arms: RVU120 + ruxolitinib

SUMMARY:
The objective of this clinical trial is to evaluate the efficacy (how well the drug works), safety, pharmacokinetics (PK), and pharmacodynamics (PD) of the study drug, RVU120, in treating adult patients with intermediate or high-risk, primary or secondary myelofibrosis. RVU120 will be given as a single agent or in combination with ruxolitinib.

DETAILED DESCRIPTION:
The study schedule consists of a screening period up to 28 days, a 21-day treatment period, an end of treatment visit (30 days) and a 1-year follow-up where participants will be contacted every 3 months for assessment. Study duration for each participant will vary depending on the number of 21-day treatment cycles received. The study is open to participants aged ≥18 years with intermediate or high-risk, primary or secondary MF who have been previously treated, are ineligible for, or had a suboptimal response to JAK inhibitor therapy. Participants must have adequate organ function (kidney, liver) and no history of hematopoietic stem cell transplant. Participants may withdraw from the study at any time at their own request or may be withdrawn at any time at the discretion of the Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Diagnosis of Primary or Secondary myelofibrosis (MF) according to the revised World Health Organization (WHO) criteria (Arber 2022).
3. Intermediate or high-risk disease.
4. Resistant or refractory to prior Janus kinase (JAK) inhibitor treatment or ineligible for JAK inhibitor treatment in the opinion of the investigator; or Suboptimal response to JAK inhibitor treatment. Note: a suboptimal response to JAK inhibitor treatment is defined as spleen size increase by palpation >25% after the first 3 months of treatment with a JAK inhibitor or persistent splenomegaly (spleen volume of >450 cm3) after at least 6 months of JAK inhibitor treatment and presence of 1 symptom score ≥5 or 2 symptom scores ≥3, new or persistent red blood cell (RBC) transfusion dependence; or may include participants naïve to previous treatment with JAK inhibitor.
5. Measurable splenomegaly as demonstrated by palpable spleen measuring ≥5 cm below the left costal margin. The edge of the spleen should be measured from the mid-clavicular line on the left side of the abdomen to the point of greatest splenic protrusion; or spleen volume of ≥450 cm3 measured by magnetic resonance imaging(MRI) or computed tomography (CT).
6. Active symptoms of MF as demonstrated by a symptom score of at least 5 points (on a 0 to 10 scale) on at least one of the symptoms or a score of 3 or greater on at least 2 of the following symptoms: night sweats, itchiness, abdominal discomfort, pain under ribs on left side, early satiety, bone or muscle pain, and inactivity.
7. Eastern Cooperative Oncology Group (ECOG) performance score 0-2.
8. Adequate hematologic function defined as:

   1. absolute neutrophil count (ANC) ≥1.0 × 109/L (without growth factor support)
   2. platelet count ≥50 × 109/L (Cohort 2 and Cohort 3 only)
9. Adequate renal function defined as calculated or measured creatinine clearance (CrCl) of ≥30 mL/minute using the formula of Cockcroft and Gault (see Section 15).
10. Adequate liver function defined as (a) aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 × upper limit of normal (ULN); (b) alkaline phosphatase (ALP) ≤2 × ULN (ALP ≤5 × ULN for participants with isozymes specific to bone); (c) bilirubin <2 × ULN or bilirubin ≤3 × ULN if due to Gilbert's disease.

Exclusion Criteria:

Each participant must not meet any of the following:

1. Peripheral blood blast count of ≥10% or bone marrow blast count of ≥10%.
2. Prior history of hematopoietic stem cell transplant.
3. Participation in any other study in which receipt of an investigational new drug occurred within 4 weeks prior to Cycle 1 Day 1.
4. Active known second malignancy with the exception of any of the following:

   1. Adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or in situ cervical cancer
   2. Adequately treated Stage I cancer from which the participant is currently in remission and has been in remission for ≥2 years
   3. Low-risk prostate cancer with a Gleason score <7 and a prostate-specific antigen (PSA) level <10 ng/mL
   4. Any other cancer from which the participant has been disease-free for ≥3 years.
5. Known or suspected allergy to RVU120 or RUX.
6. Impairment of gastrointestinal function or gastrointestinal disease
7. Major surgical procedure or significant traumatic injury within 28 days Placement of a vascular access device or minor surgery is permitted within 14 days before Cycle 1 Day 1 (provided that the wound has healed).
8. Ongoing systemic infection requiring antibiotic, antiviral, or antifungal treatment. Note: prophylactic treatment is allowed.
9. Significant cardiac dysfunction defined as myocardial infarction within 12 months of Cycle 1 Day 1, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled dysrhythmias, poorly controlled angina (Section 17), or left ventricular ejection fraction (LVEF) <40% as per echocardiography or multiple gated acquisition (MUGA) scan.
10. Taking any medications, herbal supplements, or other substances (including smoking) that are known to be strong inhibitors or moderate/strong inducers or sensitive substrates of CYP1A2, within less than 5 half-lives prior to Cycle 1 Day 1.
11. History of ventricular arrhythmia, or QTc ≥470 millisecond (Bazett's formula).
12. Known active human immunodeficiency virus (HIV) infection
13. Current active liver disease from any cause
14. Pregnant or lactating females.
15. Any other prior or current medical or psychiatric condition, intercurrent illness, surgical history, physical or electrocardiogram (ECG) findings, laboratory abnormalities, or extenuating circumstance (e.g., alcohol or drug addiction) that, in the Investigator's opinion, could jeopardize participant safety or interfere with the objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the number of participants with a response (anti-cancer activity) to RVU120 when administered as a single agent or in combination with ruxolitinib | 12 months
  The proportion of participants with spleen volume reduction (SVR) of ≥35% after 24 weeks of study treatment evaluated by magnetic resonance imaging (MRI) or computed tomography (CT)

SECONDARY OUTCOMES:
To further evaluate the number of participants having a response (anti-cancer activity and/or clinical benefit) to RVU120 when administered as a single agent or in combination with ruxolitinib | 12 months
  The proportion of participants with ≥1 Grade bone marrow fibrosis improvement after 24 weeks of study treatment
Duration of spleen response | 12 months
  Assessed as the time from initial SVR of ≥35% by MRI/CT until disease progression or death, whichever occurs first
Number of participants with leukemic transformation | 12 months
  Assessed as the proportion of participants with bone marrow blast counts of at least 20%, or peripheral blast counts of at least 20% lasting 2 weeks
Number of participants with hematological (clinical) improvement | 12 months
  Assessed as the proportion of participants with hematological (clinical) improvement as defined by International Working Group (IWG) Consensus Criteria (see Tefferi et al., 2006 for further details)
Progression-Free Survival (PFS) | 12 months
  Assessed as time from the time from first treatment to the first occurrence of disease progression or death
Overall Survival (OS) | 12 months
  Assessed as time from the time from first treatment to death
Incidence and severity of adverse events (AEs) | 12 months
  Assessed as the number and grade of adverse events assessed by CTCAE v5.0
Change in symptom burden | Baseline and week 24
  Assessed as the proportion of participants achieving at least a 50% reduction in symptom burden after 24 weeks of commencing study treatment as assessed by the Total Symptom Score (TSS) using the Myelofibrosis Symptom Assessment Form (MFSAF). Each item is rated on a scale from 0 (Absent) to 10 (Worst Imaginable).
Absolute change in TSS from baseline | Baseline and week 24
  Assessed as the number of participants with absolute change in Total Symptom Score (TSS) from baseline assessed using the Myelofibrosis Symptom Assessment Form (MFSAF). Each item is rated on a scale from 0 (Absent) to 10 (Worst Imaginable).

CONTACTS AND LOCATIONS:
Locations (18):
- Italy (5):
  - Policlinico Sant'Orsola-Malpighi, Bologna
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, Brescia
  - Azienda Ospedaliero Universitaria Policlinico "G. Rodolico - San Marco", Catania
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l., Meldola
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
- Poland (13):
  - Wojewódzki Szpital Specjalistyczny w Białej Podlaskiej, Biała Podlaska
  - Szpital Uniwersytecki nr 2 im. dr Jana Biziela, Bydgoszcz
  - M2M Med. Sp. z o.o. Sp. j., Chorzów
  - Centrum Wsparcia Badań Klinicznych UCK Ośrodek Badań Klinicznych Wczesnych Faz, Gdansk
  - Pratia Hematologia Sp. z o.o., Katowice
  - Świętokrzyskie Centrum Onkologii Samodzielny Publiczny Zakład Opieki Zdrowotnej, Kielce
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Krakow
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 w Lublinie, Lublin
  - Wojewódzki Szpital Zespolony im. L. Rydygiera w Toruniu, Torun
  - Lux Med Onkologia Sp. z o.o., Warsaw
  - Wojskowy Instytut Medyczny Państwowy Instytut Badawczy, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu, Wroclaw
  - Szpital Uniwersytecki Imienia Karola Marcinkowskiego w Zielonej Gorze Sp. z o. o., Zielona Góra

IPD SHARING:
Plan to Share IPD: No